CLINICAL TRIAL: NCT05734924
Title: Adding Low Frequancy High Intensty Magnetic Therapy to Cervical Stabilization Exercises in Cervical Spondylosis
Brief Title: Magnetic Therapy and Cervical Stabilization Exercises in Cervical Spondylosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Alzahraa Fekry Morshed, Assistant Lecturer, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003846
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cervical Spondylosis
Keywords: Cervical Spondylosis - magnetic therapy
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Intervention Model Description: The selected patients will be randomly assigned into two equal groups study group (GI), and control group (GII). The study group (GI) will receive low Frequency High Intensity magnetic therapy in addition to cervical stabilization exercise protocol . The control group (GII) will receive sham magnetic therapy in addition to, cervical stabilization exercise protocol.
Who Masked: Participant
Masking Description: The patients in control group will receive sham magnetic therapy in addition to, cervical stabilization exercise protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): The patient in this group will received low Frequency High Intensity magnetic therapy with frequency 50 Hz and high intensity 60mT for 30 minutes /session, treatment will be conducted for 3times/week for five weeks combined with cervical stabilization exercise protocol
  Interventions: Device: low Frequency High Intensity magnetic therapy
- control group (Sham Comparator): The patient in this group will sham magnetic therapy in addition to, cervical stabilization exercise protocol; treatment will conduct for 3 times/ week for five weeks.
  Interventions: Device: low Frequency High Intensity magnetic therapy

INTERVENTIONS:
Device: low Frequency High Intensity magnetic therapy — low Frequency High Intensity magnetic therapy with frequency 50 Hz and high intensity 60mT

SUMMARY:
The purposes of this study are to Investigate adding low frequency high intensity magnetic therapy to cervical stabilization exercises on pain intensity, function, ROM, cervical endurance, and cervical proprioception errors in patients with cervical spondylosis.

DETAILED DESCRIPTION:
Cervical spondylosis is a chronic degenerative process of the cervical spine. Pain in the neck and/or arms, neck stiffness, and headaches are the usual symptoms of cervical spondylosis . Low frequency high intensity magnetic therapy causes short term immediate effect in the relieve pain and improve function in patients with cervical spondylosis . Cervical stabilization causes decrease in neck pain and neck disability as well as a significant increase in cervical muscle endurance and cervical range of motion after the intervention. It also demonstrates a more ideal upper body posture and improved cervical proprioception. In the present study, therefore, we aimed to investigate adding low frequency high intensity magnetic therapy to CSE on management of cervical spondylosis. This study will be a benefit in the physical therapy field and may guide rehabilitation programs of physical therapy towards better results through decreasing time needed to perform activity of daily living, decreasing dependency and making patient an active member in society.

ELIGIBILITY:
Inclusion Criteria:

* Eighty Cervical spondylosis patients from both sexes will be participated in this study.
* The patients' ages will be ranged from 30-45 years to prevent aging process.
* X-ray evidence of cervical spondylosis (osteophyte formation, intervertebral disc height narrowing and vertebral end-plate sclerosis) .
* The presence of chronic neck pain (more than 3 months).
* Limited mobility in the cervical spine.

Exclusion Criteria:

* The following patients will be excluded from the study patients with:

  * History of cervical injury of trauma.
  * Cervical myelopathy.
  * Inflammatory arthritis involving cervical spine.
  * Tumor or infection involving cervical spine.
  * Vertebrobasilar artery insufficiency.
  * Neurologic disease (e.g. multiple sclerosis, Parkinson's disease, syringomyelia).
  * Congenital anomalies involving cervical spine.
  * Diabetes mellitus.
  * Vestibular system impairments.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of Endurance of deep neck flexor muscle by the stabilizer | Baseline
  Neck muscles endurance test will assess using the stabilizer. Subjects laid hook-lying position on a therapy table with a neutral neck position where their head and neck will be lined up and straight.
  The pressure sensor of the stabilizer will placed underneath the neck. Subjects will instructed to nod their head gently as if saying 'yes' without using the neck motions which may substitute the sternocleidomastoid muscle so that the pressure sensor will measured 2 mmHg above baseline.
  The testing will ranged from 20 mmHg to 30 mmHg and the pressure should maintain for the 10 seconds in each 2 mmHg without resting in muscle endurance test. Record the number of times a subject will hold the pressure level .

SECONDARY OUTCOMES:
Assessment of pain pressure threshold (PPT) assessment by using pressure algometer | Baseline
  A PPT measurement will be obtained in the same order for all patients. The pressure will applied with 0.785 cm2 rubber tip at tolerable level of the patient at the site of measurement.
  The measurement will be at the mid-belly of upper fiber of trapezius muscles at both sides.
  The tip of the algometer will position on this specific point. By pushing the algometer, the force will applied to the mid belly of trapezius gradually will increased.
  The patients will not allowed to see the algometer display in any moment, and, as soon as the volunteers experience a painful sensation, they say "stop", the algometer will immediately release and the force (in Kpa) will read from the display.
  A PPT will measure three times per patient on each site and the average will be calculated and will be used for analysis
Assessment of pain and function using Neck disability index (NDI): | Baseline
  The NDI will be scored as a raw score or doubled and expressed as a percent . Each section will be scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.
  Points will sum to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability

CONTACTS AND LOCATIONS:
Overall Officials: Al zahraa F Morshed, MSC, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akkan H, Gelecek N. The effect of stabilization exercise training on pain and functional status in patients with cervical radiculopathy. J Back Musculoskelet Rehabil. 2018;31(2):247-252. doi: 10.3233/BMR-169583. PMID 28946516